CLINICAL TRIAL: NCT03453970
Title: Effectiveness of a Diabetes Education Program Based on Tailored Interventions in the Andalusian Public Health and Social System (Edep-Ti Study).
Brief Title: Effectiveness of a Diabetes Education Program Based on Tailored Interventions (Edep-Ti Study)
Acronym: Edep-Ti
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, JOSE MIGUEL MORALES ASENCIO, Professor, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AP-0005-2015 / PI14-01127
Record Dates: First submitted 2018-01-17; First posted 2018-03-05 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: patient education; self-care; Controlled Trial
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic Education Program (Experimental): The program is based on adapted interventions and will consist of the following phases:
  Phase I: Identification of self-care needs in Diabetes Mellitus through the EBADE questionnaire. This instrument will identify the needs grouped by constructs of the theory of planned behavior (behavioral beliefs, subjective norm, behaviors of perceived control and behavioral intention).
  Phase II: Application of interventions adapted according to the behavioral mediator who encounters barriers. The interventions will be applied both in the face-to-face and telephone modality, using the Nursing Intervention Classification and their respective activities.
  Phase III: measurement of the clinical variables and reported by the patients described in the objectives.
  Interventions: Behavioral: Therapeutic Education Program
- Usual Care (No Intervention): The conventional intervention consists of the usual care that is followed in the nursing consultations in primary care to patients with type 2 DM, based on the recommendations of the Clinical Practice Guide of the National Health System

INTERVENTIONS:
Behavioral: Therapeutic Education Program — The total duration of the program will be 12 weeks with a maximum of 6 sessions of 30 minutes each. In the first session, through the EBADE questionnaire, the needs will be identified by grouping them by the 4 constructs of the theory of planned behavior (behavioral beliefs, subjective norm, behaviors of perceived control and behavioral intention). The interventions and the number of sessions will be adapted depending on the areas identified with barriers. These interventions will be applied in both face-to-face and telephone modalities, using the Nursing Intervention Classification and their respective activities. The interventions will be carried out by nurses who have previously received training on the proposed program. Follow-ups will be carried out every 15 days.
  Arms: Therapeutic Education Program

SUMMARY:
GOALS:

PRIMARY:

1. Analyze the overall impact of the proposed diabetes education program on metabolic control (HbA1c) and modifiable cardiovascular risk factors (lipid profile and blood pressure).

   SECONDARY:
2. Evaluate the effectiveness of the program on smoking habits and body mass index (weight, height).
3. Analyze the impact of the program on the quality of life related to health.
4. Check the effect on lifestyles: compliance levels of physical exercise and adherence to diet mediterranean.

DESIGN: Cluster randomized controlled trial

DETAILED DESCRIPTION:
The reference population will be patients with a diagnosis of diabetes mellitus in treatment with oral antidiabetics, excluding the insulinized patients. They will then be randomly assigned by cluster, to the intervention group (individual education) or control (usual care) in the context of each health center participating in the project. After randomization centers, all professionals who decide to cooperate receive a training process on methodology for measuring results (clinical and questionnaire variables), while assigned to the experimental intervention, will also receive training on how to carry out the program of diabetologic education proposed. The follow-up period for both groups is 18 months obtained as clinical determinations: glycosylated hemoglobin (metabolic control), blood pressure, lipid profile, smoking and BMI; and as results reported by the patient through questionnaires: quality of life related to health, level of physical activity performed or adherence to the Mediterranean diet.

ELIGIBILITY:
Inclusion Criteria:

- Patients with Type II Diabetes Mellitus diagnosed <10 years and classified in a computerized clinical history with poor metabolic control (HbA1c> 7% or BMI > 27.5) and in treatment with oral antidiabetics.

Exclusion Criteria:

* Diabetes Mellitus type 1
* Insulinized patients.
* Patients who have received some type of structured educational intervention in the last year according to the data obtained in their clinical history.
* Patients with some type of sensory or mental disability.
* Gestational diabetes.
* Patients with age equal to or greater than 75 years of age or minors.
* Patients with inability to travel to their Health Center.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change from basal glycosylated hemoglobin (HbA1c) at 6 months, change from basal HbA1c at 12 months and change from basal HbA1c at 18 months | 0,6,12 and18 months
  Determination of HbA1c measured as a percentage
Lipidic profile: change from basal total cholesterol (TC) at 6 months, change from total basal cholesterol at 12 months and change from total basal cholesterol at 18 months. | 0,6,12 and18 months
  Determination of total cholesterol (TC) values measured in milligrams per deciliter (mg/dl).
Lipidic profile: change from baseline LDL cholesterol (LDLc) at 6 months, change from baseline LDLc at 12 months and change from baseline LDL cholesterol at 18 months. | 0,6,12 and18 months
  Determination of LDLc measured in milligrams per deciliter (mg/dl).
Lipidic profile:change from basal triglyceride (TG) levels at 6 months, change from basal TG levels at 12 months and change from baseline TG levels at 18 months. | 0,6,12 and18 months
  Determination of TG measured in milligrams per deciliter (mg/dl).
Change from baseline systolic blood pressure (SBP) at 6 months, change from baseline systolic blood pressure at 12 months and change from baseline systolic blood pressure at 18 months. | 0,6,12 and18 months
  Determination of systolic blood pressure measured in millimeters of mercury (mm / Hg), average of 2 determinations.
Change from baseline diastolic blood pressure (DBP) at 6 months, change from baseline diastolic blood pressure at 12 months and change from baseline diastolic blood pressure at 18 months. | 0,6,12 and18 months
  Determination of diastolic blood pressure measured in millimeters of mercury (mm / Hg), average of 2 determinations.

SECONDARY OUTCOMES:
Development in smoking habits | 0,6,12 and18 months
  Number of cigarettes consumed per day on average (measured at 0,6,12 and 18 months)
Smoking rate | 0,6,12 and18 months
  Percentage of smokers of the total of the participants (measured at 0,6,12 and 18 months).
Change from baseline weight at 6 months, change from baseline weight at 12 months and change from baseline weight at 18 months. | 0,6,12 and18 months
  Determination of the body mass index calculated as the weight measured in kilograms (kg) divided by the height measured in meters squared (weight / height2) (Kg /m2) (measured at 0,6,12 and 18 months).
Change in the quality of life related to health (HRQoL) from the baseline determination at 6 months, change in the HRQoL from the baseline determination at 12 months and change in the HRQoL from the baseline determination at 18 months. | 0,6,12 and18 months
  The Diabetes Quality of Life Questionnaire EuroQol-5D (EQ-5D) in a Spanish version will be implemented at 0, 6, 12 and 18 months. With this questionnaire the individual himself assesses his health status, first in levels of severity (1-without problems, 2-some problems or moderate problems and 3-serious problems) by health dimensions (mobility, personal care, daily activities, pain/discomfort and anxiety / depression). The combination of the values of all dimensions generates 5-digit numbers, with 243 combinations of possible health states. A second part of the questionnaire includes a vertical analog visual scale ranging from 0 (worst imaginable health status) to 100 (best imaginable health status). In it, the individual must mark the point in the vertical line that best reflects his or her subjective assessment of their overall health status.
Change from the basal level of physical activity to 6 months, change from the basal level of physical activity to 12 months and change from the basal level of physical activity to 18 months. | 0,6,12 and18 months
  The International Physical Activity Questionnaire (IPAQ short version) will be implemented at 0, 6, 12 and 18 months. The IPAQ questionnaire in its short version is self-administered and consists of 7 questions that provide information on the time spent doing physical activities of moderate and vigorous intensity, separating time spent walking and time spent in a more passive state. Individuals can be classified into: low level of activity, moderate level (there are 3 criteria to classify a person as active) and high level of activity (there are 2 criteria to classify a person as very active).
Change from the baseline level of adherence to the diet at 6 months, change from the baseline level of adherence to the diet at 12 months and change from the baseline level of adherence to the diet at 18 months. | 0,6,12 and18 months
  The Questionnaire of Adherence to the Mediterranean Diet will be implemented at 0, 6, 12 and 18 months. It is a self-administered questionnaire consisting of 14 segments dedicated to eating habits. To estimate the results, the value 1 is assigned to each segment with an affirmative response and 0 to each segment with a non compliant response. From the sum of the values obtained, the degree of adherence is determined, establishing two levels, so that if the total score is greater than or equal to 9 it is considered a diet with a good level of adherence and if the total sum is lower of 9 the diet is considered to be of a low adherence.

OTHER OUTCOMES:
Change from the initial assessment of barriers to self-care at 6 months, change from the initial assessment of barriers to self-care at 12 months and change from the initial assessment of barriers to self-care at 18 months | 0,6,12 and18 months
  The questionnaire of evaluation of self-care barriers in diabetes (EBADE questionnaire) will be implemented at 0, 6, 12 and 18 months. This questionnaire consists of 15 items and 4 structured dimensions according to the Theory of Planned Behavior (behavioral beliefs, subjective norm, behavior of perceived control and behavioral intention), with a minimum score of 15 and a maximum of 105, higher score means better level of self-care behavior. The segments include questions related to diet, physical activity, medication, foot care, control of complications and accessibility to the health system.
Participation in the program | 18 months
  Number of sessions attended

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Caro Bautista, PhD, Principal Investigator — University of Malaga
Locations (1):
- Public Health Service of Andalucía, Málaga, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aguilar Diosdado M et al. II Plan Integral de Diabetes de Andalucía: 2009-2013. Sevilla: Consejería de Salud,2009
- [Background] American Diabetes Association. Standars of Medical Care in Diabetes. Diabetes Care. 2015; 38(Suppl. 1):S1-2. DOI: 10.2337/dc15-S001
- [Background] Andersson C, van Gaal L, Caterson ID, Weeke P, James WP, Coutinho W, Finer N, Sharma AM, Maggioni AP, Torp-Pedersen C. Relationship between HbA1c levels and risk of cardiovascular adverse outcomes and all-cause mortality in overweight and obese cardiovascular high-risk women and men with type 2 diabetes. Diabetologia. 2012 Sep;55(9):2348-55. doi: 10.1007/s00125-012-2584-3. Epub 2012 May 26. PMID 22638548
- [Background] Ajzen I. The theory of planned behavior. Organ. Behav. Hum. Decis. Process. 1991; 50(2):179-211.
- [Background] Blackberry ID, Furler JS, Best JD, Chondros P, Vale M, Walker C, Dunning T, Segal L, Dunbar J, Audehm R, Liew D, Young D. Effectiveness of general practice based, practice nurse led telephone coaching on glycaemic control of type 2 diabetes: the Patient Engagement and Coaching for Health (PEACH) pragmatic cluster randomised controlled trial. BMJ. 2013 Sep 18;347:f5272. doi: 10.1136/bmj.f5272. PMID 24048296
- [Background] Campbell M, Fitzpatrick R, Haines A, Kinmonth AL, Sandercock P, Spiegelhalter D, Tyrer P. Framework for design and evaluation of complex interventions to improve health. BMJ. 2000 Sep 16;321(7262):694-6. doi: 10.1136/bmj.321.7262.694. No abstract available. PMID 10987780
- [Background] Carnethon MR, De Chavez PJ, Biggs ML, Lewis CE, Pankow JS, Bertoni AG, Golden SH, Liu K, Mukamal KJ, Campbell-Jenkins B, Dyer AR. Association of weight status with mortality in adults with incident diabetes. JAMA. 2012 Aug 8;308(6):581-90. doi: 10.1001/jama.2012.9282. PMID 22871870
- [Background] Cardenas-Valladolid J, Salinero-Fort MA, Gomez-Campelo P, de Burgos-Lunar C, Abanades-Herranz JC, Arnal-Selfa R, Andres AL. Effectiveness of standardized Nursing Care Plans in health outcomes in patients with type 2 Diabetes Mellitus: a two-year prospective follow-up study. PLoS One. 2012;7(8):e43870. doi: 10.1371/journal.pone.0043870. Epub 2012 Aug 27. PMID 22952794
- [Background] Caro-Bautista J, Martin-Santos FJ, Villa-Estrada F, Morilla-Herrera JC, Cuevas-Fernandez-Gallego M, Morales-Asencio JM. Using qualitative methods in developing an instrument to identify barriers to self-care among persons with type 2 diabetes mellitus. J Clin Nurs. 2015 Apr;24(7-8):1024-37. doi: 10.1111/jocn.12740. Epub 2014 Dec 19. PMID 25523621
- [Background] Caro-Bautista J, Martin-Santos FJ, Morales-Asencio JM. Systematic review of the psychometric properties and theoretical grounding of instruments evaluating self-care in people with type 2 diabetes mellitus. J Adv Nurs. 2014 Jun;70(6):1209-27. doi: 10.1111/jan.12298. Epub 2013 Nov 17. PMID 24237156
- [Background] Cassimatis M, Kavanagh DJ. Effects of type 2 diabetes behavioural telehealth interventions on glycaemic control and adherence: a systematic review. J Telemed Telecare. 2012 Dec;18(8):447-50. doi: 10.1258/jtt.2012.gth105. Epub 2012 Dec 3. PMID 23209266
- [Background] Claydon-Platt K, Manias E, Dunning T. The barriers and facilitators people with diabetes from a nonEnglish speaking background experience when managing their medications: a qualitative study. J Clin Nurs. 2014 Aug;23(15-16):2234-46. doi: 10.1111/jocn.12501. Epub 2013 Dec 26. PMID 24372586
- [Background] Deakin T, McShane CE, Cade JE, Williams RD. Group based training for self-management strategies in people with type 2 diabetes mellitus. Cochrane Database Syst Rev. 2005 Apr 18;(2):CD003417. doi: 10.1002/14651858.CD003417.pub2. PMID 15846663
- [Background] Debussche X, Collin F, Fianu A, Balcou-Debussche M, Fouet-Rosiers I, Koleck M, Favier F. Structured self-management education maintained over two years in insufficiently controlled type 2 diabetes patients: the ERMIES randomised trial in Reunion Island. Cardiovasc Diabetol. 2012 Aug 2;11:91. doi: 10.1186/1475-2840-11-91. PMID 22856504
- [Background] Didarloo AR, Shojaeizadeh D, Gharaaghaji Asl R, Habibzadeh H, Niknami Sh, Pourali R. Prediction of Self-Management Behavior among Iranian Women with Type 2 Diabetes: Application of the Theory of Reasoned Action along with Self-Efficacy (ETRA). Iran Red Crescent Med J. 2012 Feb;14(2):86-95. Epub 2012 Feb 1. PMID 22737561
- [Background] Duke SA, Colagiuri S, Colagiuri R. Individual patient education for people with type 2 diabetes mellitus. Cochrane Database Syst Rev. 2009 Jan 21;2009(1):CD005268. doi: 10.1002/14651858.CD005268.pub2. PMID 19160249
- [Background] Drewelow E, Wollny A, Pentzek M, Immecke J, Lambrecht S, Wilm S, Schluckebier I, Loscher S, Wegscheider K, Altiner A. Improvement of primary health care of patients with poorly regulated diabetes mellitus type 2 using shared decision-making--the DEBATE trial. BMC Fam Pract. 2012 Aug 22;13:88. doi: 10.1186/1471-2296-13-88. PMID 22913642
- [Background] Edelman D, Dolor RJ, Coffman CJ, Pereira KC, Granger BB, Lindquist JH, Neary AM, Harris AJ, Bosworth HB. Nurse-led behavioral management of diabetes and hypertension in community practices: a randomized trial. J Gen Intern Med. 2015 May;30(5):626-33. doi: 10.1007/s11606-014-3154-9. Epub 2015 Jan 8. PMID 25567758
- [Background] Espelt A, Kunst AE, Palencia L, Gnavi R, Borrell C. Twenty years of socio-economic inequalities in type 2 diabetes mellitus prevalence in Spain, 1987-2006. Eur J Public Health. 2012 Dec;22(6):765-71. doi: 10.1093/eurpub/ckr158. Epub 2011 Oct 29. PMID 22037802
- [Background] Fu AZ, Qiu Y, Radican L, Yin DD, Mavros P. Impact of concurrent macrovascular co-morbidities on healthcare utilization in patients with type 2 diabetes in Europe: a matched study. Diabetes Obes Metab. 2010 Jul;12(7):631-7. doi: 10.1111/j.1463-1326.2010.01200.x. PMID 20590738
- [Background] Gabbay RA, Anel-Tiangco RM, Dellasega C, Mauger DT, Adelman A, Van Horn DH. Diabetes nurse case management and motivational interviewing for change (DYNAMIC): results of a 2-year randomized controlled pragmatic trial. J Diabetes. 2013 Sep;5(3):349-57. doi: 10.1111/1753-0407.12030. Epub 2013 May 28. PMID 23368423
- [Background] Gil Montalban E, Zorrilla Torras B, Ortiz Marron H, Martinez Cortes M, Donoso Navarro E, Nogales Aguado P, de la Calle Blasco H, Medrano Albero MJ, Cuadrado Gamarra I. [Prevalence of diabetes mellitus and cardiovascular risk factors in the adult population of the autonomous region of Madrid (Spain): the PREDIMERC study]. Gac Sanit. 2010 May-Jun;24(3):233-40. doi: 10.1016/j.gaceta.2010.01.010. Epub 2010 Apr 8. Spanish. PMID 20381212
- [Background] Gomis R, Artola S, Conthe P, Vidal J, Casamor R, Font B; investigadores del Grupo de Estudio OBEDIA. [Prevalence of type 2 diabetes mellitus in overweight or obese outpatients in Spain. OBEDIA Study]. Med Clin (Barc). 2014 Jun 6;142(11):485-92. doi: 10.1016/j.medcli.2013.03.013. Epub 2013 May 15. Spanish. PMID 23683969
- [Background] Grau M, Elosua R, Cabrera de Leon A, Guembe MJ, Baena-Diez JM, Vega Alonso T, Javier Felix F, Zorrilla B, Rigo F, Lapetra J, Gavrila D, Segura A, Sanz H, Fernandez-Berges D, Fito M, Marrugat J. [Cardiovascular risk factors in Spain in the first decade of the 21st Century, a pooled analysis with individual data from 11 population-based studies: the DARIOS study]. Rev Esp Cardiol. 2011 Apr;64(4):295-304. doi: 10.1016/j.recesp.2010.11.005. Spanish. PMID 21397375
- [Background] Grupo de trabajo de la Guía de Práctica Clínica sobre Diabetes tipo 2. Guía de Práctica Clínica sobre Diabetes tipo 2. Madrid: Plan Nacional para el SNS del MSC. Agencia de Evaluación de Tecnologías Sanitarias del País Vasco; 2008. Guías de Práctica Clínica en el SNS: OSTEBA No 2006/08.
- [Background] Heinrich E, de Nooijer J, Schaper NC, Schoonus-Spit MH, Janssen MA, de Vries NK. Evaluation of the web-based Diabetes Interactive Education Programme (DIEP) for patients with type 2 diabetes. Patient Educ Couns. 2012 Feb;86(2):172-8. doi: 10.1016/j.pec.2011.04.032. Epub 2011 May 26. PMID 21616626
- [Background] International Standards for Diabetes Education [Internet]. [citado 12 de febrero de 2012]. Recuperado a partir de: http://www.idf.org/node/1684.
- [Background] Inzucchi SE, Bergenstal RM, Buse JB, Diamant M, Ferrannini E, Nauck M, Peters AL, Tsapas A, Wender R, Matthews DR. Management of hyperglycaemia in type 2 diabetes: a patient-centered approach. Position statement of the American Diabetes Association (ADA) and the European Association for the Study of Diabetes (EASD). Diabetologia. 2012 Jun;55(6):1577-96. doi: 10.1007/s00125-012-2534-0. Epub 2012 Apr 20. No abstract available. PMID 22526604
- [Background] Jimenez Mejias E, Olvera Porcel MC, Amezcua Prieto C, Olmedo-Requena R, Martinez Ruiz V, Jimenez Moleon JJ. [Effect of age on the prevalence of diabetes mellitus in Spain between 2001 and 2012]. Nutr Hosp. 2014 Jun 1;29(6):1335-8. doi: 10.3305/nh.2014.29.6.7327. Spanish. PMID 24972471
- [Background] Khunti K, Gray LJ, Skinner T, Carey ME, Realf K, Dallosso H, Fisher H, Campbell M, Heller S, Davies MJ. Effectiveness of a diabetes education and self management programme (DESMOND) for people with newly diagnosed type 2 diabetes mellitus: three year follow-up of a cluster randomised controlled trial in primary care. BMJ. 2012 Apr 26;344:e2333. doi: 10.1136/bmj.e2333. PMID 22539172
- [Background] Lakerveld J, Bot SD, Chinapaw MJ, Knol DL, de Vet HC, Nijpels G. Measuring pathways towards a healthier lifestyle in the Hoorn Prevention Study: the Determinants of Lifestyle Behavior Questionnaire (DLBQ). Patient Educ Couns. 2011 Nov;85(2):e53-8. doi: 10.1016/j.pec.2011.01.014. Epub 2011 Feb 5. PMID 21296535
- [Background] Li W, Katzmarzyk PT, Horswell R, Zhang Y, Zhao W, Wang Y, Johnson J, Hu G. Body mass index and stroke risk among patients with type 2 diabetes mellitus. Stroke. 2015 Jan;46(1):164-9. doi: 10.1161/STROKEAHA.114.006718. Epub 2014 Dec 2. PMID 25468880
- [Background] Mc Hugh S, O'Mullane M, Perry IJ, Bradley C. Barriers to, and facilitators in, introducing integrated diabetes care in Ireland: a qualitative study of views in general practice. BMJ Open. 2013 Aug 19;3(8):e003217. doi: 10.1136/bmjopen-2013-003217. PMID 23959754
- [Background] Millan M. [Quality-of-life questionnaire designed for diabetes mellitus (EsDQOL)]. Aten Primaria. 2002 May 15;29(8):517-21. doi: 10.1016/s0212-6567(02)70623-9. No abstract available. Spanish. PMID 12031227
- [Background] Raaijmakers LG, Hamers FJ, Martens MK, Bagchus C, de Vries NK, Kremers SP. Perceived facilitators and barriers in diabetes care: a qualitative study among health care professionals in the Netherlands. BMC Fam Pract. 2013 Aug 10;14:114. doi: 10.1186/1471-2296-14-114. PMID 23937325
- [Background] Radhakrishnan K. The efficacy of tailored interventions for self-management outcomes of type 2 diabetes, hypertension or heart disease: a systematic review. J Adv Nurs. 2012 Mar;68(3):496-510. doi: 10.1111/j.1365-2648.2011.05860.x. Epub 2011 Oct 20. PMID 22010971
- [Background] Roman-Viñas B, Serra-Majem L, Hagströmer M, Ribas-Barba L, Sjöström M, Segura-Cardona R. International Physical Activity Questionnaire: Reliability and validity in a Spanish population. Eur. J. Sport Sci. 2010; 10(5):297-304.
- [Background] Soriguer F, Goday A, Bosch-Comas A, Bordiu E, Calle-Pascual A, Carmena R, Casamitjana R, Castano L, Castell C, Catala M, Delgado E, Franch J, Gaztambide S, Girbes J, Gomis R, Gutierrez G, Lopez-Alba A, Martinez-Larrad MT, Menendez E, Mora-Peces I, Ortega E, Pascual-Manich G, Rojo-Martinez G, Serrano-Rios M, Valdes S, Vazquez JA, Vendrell J. Prevalence of diabetes mellitus and impaired glucose regulation in Spain: the Di@bet.es Study. Diabetologia. 2012 Jan;55(1):88-93. doi: 10.1007/s00125-011-2336-9. Epub 2011 Oct 11. PMID 21987347
- [Background] Sperl-Hillen J, Beaton S, Fernandes O, Von Worley A, Vazquez-Benitez G, Parker E, Hanson A, Lavin-Tompkins J, Glasrud P, Davis H, Adams K, Parsons W, Spain CV. Comparative effectiveness of patient education methods for type 2 diabetes: a randomized controlled trial. Arch Intern Med. 2011 Dec 12;171(22):2001-10. doi: 10.1001/archinternmed.2011.507. Epub 2011 Oct 10. PMID 21986350
- [Background] Steinsbekk A, Rygg LO, Lisulo M, Rise MB, Fretheim A. Group based diabetes self-management education compared to routine treatment for people with type 2 diabetes mellitus. A systematic review with meta-analysis. BMC Health Serv Res. 2012 Jul 23;12:213. doi: 10.1186/1472-6963-12-213. PMID 22824531
- [Background] Tressler MC, Greer N, Rector TS, Ishani A, Ercan-Fang N. Factors associated with treatment success in veterans with diabetes and hyperlipidemia: a retrospective study. Diabetes Educ. 2013 Sep-Oct;39(5):664-70. doi: 10.1177/0145721713492568. Epub 2013 Jun 19. PMID 23782624
- [Background] Trichopoulou A, Costacou T, Bamia C, Trichopoulos D. Adherence to a Mediterranean diet and survival in a Greek population. N Engl J Med. 2003 Jun 26;348(26):2599-608. doi: 10.1056/NEJMoa025039. PMID 12826634
- [Background] van der Wulp I, de Leeuw JR, Gorter KJ, Rutten GE. Effectiveness of peer-led self-management coaching for patients recently diagnosed with Type 2 diabetes mellitus in primary care: a randomized controlled trial. Diabet Med. 2012 Oct;29(10):e390-7. doi: 10.1111/j.1464-5491.2012.03629.x. PMID 22414198
- [Background] Vamos EP, Harris M, Millett C, Pape UJ, Khunti K, Curcin V, Molokhia M, Majeed A. Association of systolic and diastolic blood pressure and all cause mortality in people with newly diagnosed type 2 diabetes: retrospective cohort study. BMJ. 2012 Aug 30;345:e5567. doi: 10.1136/bmj.e5567. PMID 22936794
- [Background] Whiting DR, Guariguata L, Weil C, Shaw J. IDF diabetes atlas: global estimates of the prevalence of diabetes for 2011 and 2030. Diabetes Res Clin Pract. 2011 Dec;94(3):311-21. doi: 10.1016/j.diabres.2011.10.029. Epub 2011 Nov 12. PMID 22079683
- [Background] Wilson A, O'Hare JP, Hardy A, Raymond N, Szczepura A, Crossman R, Baines D, Khunti K, Kumar S, Saravanan P; ICCD trial group. Evaluation of the clinical and cost effectiveness of intermediate care clinics for diabetes (ICCD): a multicentre cluster randomised controlled trial. PLoS One. 2014 Apr 15;9(4):e93964. doi: 10.1371/journal.pone.0093964. eCollection 2014. PMID 24736243